CLINICAL TRIAL: NCT05515939
Title: Evaluating the Utility of the "sMart" InPen Wireless-Enabled System to impRove Glycemic Control in Pediatric Type 1 Diabetes (EMPoWER Study)
Brief Title: Evaluating the InPen in Pediatric Type 1 Diabetes
Acronym: EMPoWER
Status: Active, not recruiting | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Colleen Buggs-Saxton, MD, PhD, Associate Professor of Pediatrics, Wayne State University
Other Study IDs: WSU-12-2021
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- InPen: Patients who will begin using the InPen device as per standard of care
  Interventions: Device: InPen Insulin Pen

INTERVENTIONS:
Device: InPen Insulin Pen — The InPen is a reusable smart insulin pen for people living with diabetes. The device uses Bluetooth technology to send dose information to a mobile application. The InPen can be used to deliver insulin, help calculate insulin doses, and estimate carbohydrates for meals

SUMMARY:
Type 1 Diabetes (T1D) is the most common form of diabetes affecting children, requiring lifelong administration of insulin to prevent complications. The incidence of T1D has increased more among African Americans, Hispanics, and Asian/Pacific Islanders compared to Caucasian youths in the past two decades. Despite advances in insulin delivery systems, fewer black and Hispanic children compared to white children with T1D use insulin pumps. Therefore, most minority children with T1D in urban areas require multiple daily injections (MDI) of insulin which may put them at increased risk of poor glycemic control. Although several factors contribute to worsening glycemic control in adolescents with T1D, studies have shown that missing doses of insulin at mealtimes is a major factor.

Adolescents with T1D who use MDI with a basal-bolus regimen use formulas to calculate insulin doses that involve a four-step process. The complexity of determining insulin doses contributes to inaccuracies in both timing of doses and amount of insulin given, both of which can lead to hyperglycemia and hypoglycemia.

The InPen™ Smart Insulin Pen System (Medtronics) was approved by the FDA for children of all ages with T1D in June 2020. The InPen is a Bluetooth-enabled smart insulin pen that helps with management of insulin dosing and tracking via capture of rapid-acting insulin doses and tracking of insulin in the body through the use of its companion app (free on Apple iOS and Android). The app includes a bolus calculator, which can lead to more accurate insulin dosing, which may improve glycemic control.

The specific benefits of using the InPen include the following: simplifying insulin dose calculations, administering more accurate insulin doses, tracking insulin doses to help prevent hypoglycemia, providing reminders to administer insulin, and storing data in the InPen App that can be easily shared with diabetes healthcare teams to assist with adjusting insulin doses.

The goal of this study is to determine if use of the InPen will improve glycemic control and diabetes numeracy in adolescents with uncontrolled T1D living in urban areas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 13-21 years of age (inclusive) at the time of enrollment.
2. Patients diagnosed with type 1 diabetes for more than 6 months.
3. Patients with uncontrolled T1D as defined by an elevated HbA1c > 8% within the last 3 months prior to the start of the study.
4. Patients using multiple daily injections of insulin (MDI); basal- bolus regimen requiring three or more injections per day.

   1. Basal insulin requirement: one or two dose per day of a long-acting insulin analog: insulin glargine U-100 (Lantus or Basaglar), insulin glargine U-300 (Toujeo), insulin detemir (Levemir), or insulin degludec (Tresiba).
   2. Bolus insulin requirement: three or more doses per day of a rapid-acting insulin analog: insulin lispro (Humalog or Admelog) or insulin aspart (Novolog or Fiasp).
5. Completion of basic diabetes education program within first year of diagnosis including management of hyperglycemia and hypoglycemia.
6. Patients not actively using InPen (including discontinuation of the InPen for at least 12 weeks).

Exclusion Criteria:

1. Pediatric patients with T1D with health conditions that may impact glycemic control (e.g., uncontrolled hypothyroidism or hyperthyroidism or prolonged use (more than 2 weeks) of exogenous steroids), pregnancy, language barrier, or inability to obtain informed consent from patient and/or caregiver.
2. Patients who are unable to obtain insurance approval to cover the cost for the InPen device and insulin cartridges for the InPen.
3. Patients with T1D who are allergic to Humalog and Novolog insulin analogs.
4. Patients/caregivers who are unwilling to switch to the InPen device and/or insulin cartridges required for the use of the InPen device.
5. Patients who do not own a smartphone or tablet that is compatible with the InPen App.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 13-21 years of age with Type 1 Diabetes who will be initiating treatment with the InPen insulin pen device
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline to 12 and 24 weeks (End of study)
  Change in mean hemoglobin A1c (HbA1c) among patients from baseline to 12- and 24 weeks after using the InPen device in diabetes management plan.

SECONDARY OUTCOMES:
Change in Diabetes Numeracy Test (DNT-14) | Baseline and 24 weeks (end of study)
  Assessment test designed to investigate numeracy skills in patients with diabetes
Clinical Evaluation of Treatment | 24 weeks (end of study)
  Questionnaire to assess usability, comfort with, and usefulness of the InPen and its app.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT05515939/ICF_000.pdf